CLINICAL TRIAL: NCT06646679
Title: Intelligent Segmentation Algorithm of Ultrasonic Image
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Tianzhu Liu, Principal Investigator, Tongji Hospital
Other Study IDs: Tongji Hospital102114-4
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Segmentation
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasonic imaging — Ultrasonic imaging

SUMMARY:
This project aims to enhance the performance of ultrasonic image analysis by optimizing and refining neural network algorithms, while also collecting and constructing extensive datasets relevant to ultrasonic imagery. The algorithm will be trained and evaluated in a data-driven manner, with test results facilitating accurate segmentation of regional block images and identification of characteristic ultrasonic anatomy. This approach will significantly advance the study and development of ultrasonic technology.

DETAILED DESCRIPTION:
1. Algorithm development: Develop high-performance intelligent ultrasonic image recognition and segmentation algorithms;
2. Data set: Establish ultrasound image data set, which is convenient for researchers to develop and verify algorithms;
3. Apply for patents, publish academic papers, promote and popularize technology.

ELIGIBILITY:
Inclusion Criteria:

* None.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patient undergoing an ultrasound scan, including volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2026-11-14 (Estimated)

PRIMARY OUTCOMES:
Ultrasonic image | 2 years
  Ultrasound images obtained by ultrasound scan

CONTACTS AND LOCATIONS:
Overall Officials: Mei Wei, M.D., Principal Investigator — Tongji Hospital
Locations (1):
- Tianzhu Liu, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Contact the researcher if necessary after the study is completed.